CLINICAL TRIAL: NCT03044899
Title: African Surgical Outcomes Study (ASOS): An African, Multi-centre Seven Day Evaluation of Patient Care and Clinical Outcomes for Patients Undergoing Surgery
Brief Title: African Surgical Outcomes Study (ASOS)
Acronym: ASOS
Status: Completed | Type: Observational
Sponsor: University of KwaZulu (Other)
Collaborators: Medical Research Council, South Africa (Other)
Responsible Party: Sponsor
Other Study IDs: ASOS
Record Dates: First submitted 2017-02-03; First posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Surgery; Surgery- Complications; Mortality
Keywords: Surgery; Complications; Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult surgical patients: All surgeries in adult patients
  Interventions: Procedure: All surgeries in adult patients

INTERVENTIONS:
Procedure: All surgeries in adult patients — All surgeries in adult patients

SUMMARY:
STUDY OBJECTIVE To confirm the incidence of in-hospital postoperative complications in adult surgical patients in Africa.

STUDY DESIGN Seven day, African national multi-centre prospective observational cohort study of adult (≥18 years) patients undergoing surgery. Patients will be followed up for a maximum of 30 days. We will follow the original International Surgical Outcomes Study (ISOS) study design.

The primary outcome is in-hospital postoperative complications in adult surgical patients in Africa. Secondary outcomes include in-hospital mortality and the relationship between postoperative complications and postoperative mortality.

The intention is to present a representative sample of surgical outcomes across all African countries. This study will run between February and March 2016.

DETAILED DESCRIPTION:
Research questions

Primary objective To confirm the incidence of in-hospital postoperative complications in adult surgical patients in Africa Secondary objectives

1. To confirm the rate of mortality on the day of surgery for patients undergoing surgery in Africa.
2. To confirm the in-hospital mortality rate for patients undergoing surgery in Africa.
3. To describe the relationship between postoperative complications and postoperative mortality.
4. To describe the proportional contribution of communicable, non-communicable diseases and traumatic injuries to in-hospital mortality and critical care admissions in Africa.

Methods Seven day, African national multi-centre cohort study of adult (≥18 years) patients undergoing surgery. This study will be registered on ClinicalTrials.gov.

Inclusion criteria All consecutive patients admitted to participating centres undergoing elective and non-elective surgery commencing during a seven day study cohort period with a planned overnight hospital stay following surgery. The recruitment week will run between February and March 2016.

Exclusion criteria Patients undergoing planned day-case surgery or radiological procedures not requiring anaesthesia.

Centres Our plan is to recruit as many centres as possible on an international basis and ask them to include all eligible patients in the study.

Number of centres. We plan to recruit as many centres from each country for participation. Countries are expected to contribute data from at least 10 centres. Where countries have less than 10 centres performing surgery nationally, at least 50% of the surgical centres need to contribute data to ASOS.

Number of patients Only centres which provide patient data on at least 90% of the eligible surgical cases for the recruitment week will be included in the data analysis. The selected recruitment week for a country will be decided by the National Leader.

Ethics approval The requirement for patient consent is expected to vary according to regulations of the participating nations. The national leaders will ensure ethics approval is obtained from their respective countries and centres. Centres will not be permitted to record data unless ethics approval or an equivalent waiver is in place.

This study is in effect a large scale clinical audit. We expect that in most, if not every country, that there will be no requirement for individual patient consent as all data will be anonymised and is already recorded as part of routine clinical care. This international precedent has already been set, as in the original European Surgical Outcomes Study (EuSOS), consent was waived in 27 of the 28 European countries participating, and seven of the eight ethics committees in the South African Surgical Outcomes Study (SASOS).

Data collection and collation Data will be collected in individual centres on paper case record forms (CRFs) for every patient recruited. Paper CRFs will be stored within a locked office in each centre as they will include identifiable patient data in order to allow follow-up of clinical outcomes. Data will then be pseudo-anonymised by generation of a unique numeric code and transcribed by local investigators onto an internet based electronic CRF. Each patient will only be identified on the electronic CRF by their numeric code; thus the co-ordinating study team cannot trace data back to an individual patient without contact with the local team. A participant (patient) list will be used in each centre to match identifier codes in the database to individual patients in order to record clinical outcomes and supply any missing data points. Access to the data entry system will be protected by username and password delivered during the registration process for individual local investigators. All electronic data transfer between participating centres and the co-ordinating centre will be encrypted using a secure protocol.

Where individual centres are unable to access the internet based case record form, pseudo-anonymised (coded) facsimile (fax) data transfer will be available to a secure, dedicated fax machine in the co-ordinating office. Pseudo-anonymised (coded) data may also be sent by mail to the coordinating centre if necessary.

Each centre will complete a screening log reporting the number of eligible surgical patients who had surgery during the recruitment week at the centre.

Each centre will maintain a secure trial file including a protocol, local investigator delegation log, ethics approval documentation and the patient list.

Once the local co-ordinator confirms data entry is complete for their hospital they will receive a spreadsheet of raw (un-cleaned) data, allowing further checks for data completeness and accuracy.

Dataset A realistic data set will be fundamental to the success of the investigation, and this was confirmed in the EuSOS study where nearly complete data was available on 46 000 patients, and similarly in the SASOS study. We have therefore adopted core data variables from the EuSOS, International Surgical Outcomes Study (ISOS) and SASOS studies in order to achieve the study objectives. We believe that these key data points will encourage centres to participate as there will not be an excessive burden of data collection.

Centre co-ordinators may request the addition of a limited number of data points to support additional country specific data collection and for subsequent regional analyses. All additional data points must be discussed with the co-principal investigators and if necessary the steering committee.

Centre specific data will be collected once for each hospital including: university or non-university hospital, number of hospital beds, number of operating rooms, number and level of critical care beds and details about the reimbursement status of the hospital.

An ASOS case record form (CRF) will be completed for every eligible patient who undergoes surgery during the seven day cohort period (appendix 1). Patients will be followed up until hospital discharge. This will be censored at thirty days i.e. patients will be followed up until discharge or for thirty days whichever is the shorter period.

Sample size calculation Our plan is to recruit as many centres as possible from each participating country and ask them to include all eligible patients in the study. A minimum of ten centres from any country will be required for participation (with the exception of countries which have less than 10 centres performing surgery nationally, where in this circumstance at least 50% of the surgical centres need to contribute data to ASOS). Only centres including data on at least 90% of eligible patients will be included in the data analysis. We do not have a specific sample size and statistical models will be adapted to the event rate provided by the sample recruited.

Statistical analysis Data will be presented at a national level and in the following geographical regions: Northern, Western, Central, Eastern and Southern Africa. All institutional level data will be anonymised prior to publication. Categorical variables will be described as proportions and will be compared using chi-square tests. Continuous variables will be described as mean and standard deviation if normally distributed or median and inter-quartile range if not normally distributed. Comparisons of continuous variables between groups will be performed using t-tests, one-way ANOVA or equivalent non parametric tests as appropriate. Univariate analysis will be performed to test factors associated with postoperative complications, critical care admission and in-hospital death.

Single-level and hierarchical multi-level logistic regression models will be constructed to identify factors independently associated with these outcomes and to adjust for differences in confounding factors. Factors will be entered into the models based on their univariate relation to outcome (p<0.05), biological plausibility and low rate of missing data.

Results of logistic regression will be reported as adjusted odds ratios (OR) with 95% confidence intervals. The models will be assessed through the use of sensitivity analyses to explore possible interacting factors and examine any effect on the results. A single final analysis is planned at the end of the study.

Primary outcome measure Incidence of in-hospital postoperative complications in adult surgical patients in Africa.

Secondary outcome measures

1. Rate of mortality on the day of surgery for patients undergoing surgery in Africa.
2. The in-hospital mortality rate for patients undergoing surgery in Africa.

Organisation The Steering Committee will be chaired by Bruce Biccard (BB) and Thandinkosi Madiba (TM). The study management team will be appointed by the Steering Committee and led by BB and TM. The duties of this team will include administration of all project tasks, communication between project partners (including funders, steering committee members, national and local co-ordinators, etc.), data collation and management and preparation of reports for individual study sites. The Steering Committee is responsible for the scientific conduct and consistency of the project. The Steering Committee will ensure communication between the funder(s), study management team and co-ordinators as necessary.

Country co-ordinators

Country co-ordinators will be appointed by the steering committee to lead the project within individual countries and:

* Identify local co-ordinators in participating hospitals
* Assist with translation of study paperwork as required
* Ensure distribution of research manuals, CRF and other materials
* Ensure necessary regulatory approvals are in place prior to the start date
* Ensure good communication with the participating sites in his/her country

Local co-ordinators

Local co-ordinators in individual institutions will have the following responsibilities:

* Provide leadership for the study in their institution
* Ensure all relevant regulatory approvals are in place for their institution
* Ensure adequate training of all relevant staff prior to data collection
* Supervise daily data collection and assist with problem solving
* Act as guarantor for the integrity and quality of data collected
* Ensure timely completion of CRFs
* Communicate with the relevant national coordinator

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients admitted to participating centres undergoing elective and non-elective surgery commencing during a seven day study cohort period with a planned overnight hospital stay following surgery. The recruitment week will run between February and May 2016.

Exclusion Criteria:

* Patients undergoing planned day-case surgery or radiological procedures not requiring anaesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Seven day, African national multi-centre cohort study of adult (≥18 years) patients undergoing surgery.
Sampling Method: Non-Probability Sample
Enrollment: 11422 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of in-hospital postoperative complications in adult surgical patients in Africa | In-hospital upto 30 days
  Postoperative complications

SECONDARY OUTCOMES:
Rate of mortality on the day of surgery for patients undergoing surgery in Africa | 1 day
  Mortality on the day of surgery
The in-hospital mortality rate for patients undergoing surgery in Africa | In-hospital upto 30 days
  In-hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Biccard, MD, PhD, Principal Investigator — University of KwaZulu
Locations (25):
- National Coordination Office, Algiers, Algiers Province, Algeria
- National Coordination Office, Cotonou, Cotonou, Benin
- National Coordination Office, Bujumbura, Bujumbura Mairie Province, Burundi
- National Coordination Office, Mutengene, Mutengene, Cameroon
- National Coordination Office, Kinshasa, Kinshasa City, Democratic Republic of the Congo
- National Coordination Office, Cairo, Cairo Governorate, Egypt
- National Coordination Office, Addis Ababa, Addis Ababa, Ethiopia
- National Coordination Office, Kumasi, Kumasi, Ghana
- National Coordination Office, Nairobi, Nairobi County, Kenya
- National Coordination Office, Tripoli, Tripoli, Libya
- National Coordination Office, Androhibe, Tana, Madagascar
- National Coordination Office, Bamako, Bamako, Mali
- National Coordination Office, Rose Belle, Rose Belle, Mauritius
- National Coordination Office, Windhoek, Khomas Region, Namibia
- National Coordination Office, Ibadan, Ibadan, Nigeria
- National Coordination Office, Niamey, Naimey, Niger
- National Coordination Office, Brazzaville, Brazzavile Department, Republic of the Congo
- National Coordination Office, Dakar, Dakar, Senegal
- University of Kwazulu-Natal, KwaKhangela, KwaZulu-Natal, South Africa
- National Coordination Office, Mwanza, Mwanza Region, Tanzania
- National Coordination Office, Banjul, City of Banjul, The Gambia
- National Coordination Office, Tokoin, Lomé, Togo
- National Coordination Office, Kampala, Kampala, Uganda
- National Coordination Office, Lusaka, Lusaka Province, Zambia
- National Coordination Office, Harare, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van der Merwe F, Vickery NJ, Kluyts HL, Yang D, Han Y, Munlemvo DM, Ashebir DZ, Mbwele B, Forget P, Basenero A, Youssouf C, Antwi-Kusi A, Ndonga AK, Ngumi ZWW, Elkhogia A, Omigbodun AO, Tumukunde J, Madzimbamuto FD, Gobin V, Mehyaoui R, Samateh AL, du Toit L, Madiba TE, Pearse RM, Biccard BM; African Surgical Outcomes Study (ASOS) investigators. Postoperative Outcomes Associated With Procedural Sedation Conducted by Physician and Nonphysician Anesthesia Providers: Findings From the Prospective, Observational African Surgical Outcomes Study. Anesth Analg. 2022 Aug 1;135(2):250-263. doi: 10.1213/ANE.0000000000005819. Epub 2021 Dec 28. PMID 34962901
- [Derived] Bishop D, Dyer RA, Maswime S, Rodseth RN, van Dyk D, Kluyts HL, Tumukunde JT, Madzimbamuto FD, Elkhogia AM, Ndonga AKN, Ngumi ZWW, Omigbodun AO, Amanor-Boadu SD, Zoumenou E, Basenero A, Munlemvo DM, Youssouf C, Ndayisaba G, Antwi-Kusi A, Gobin V, Forget P, Mbwele B, Ndasi H, Rakotoarison SR, Samateh AL, Mehyaoui R, Patel-Mujajati U, Sani CM, Esterhuizen TM, Madiba TE, Pearse RM, Biccard BM; ASOS investigators. Maternal and neonatal outcomes after caesarean delivery in the African Surgical Outcomes Study: a 7-day prospective observational cohort study. Lancet Glob Health. 2019 Apr;7(4):e513-e522. doi: 10.1016/S2214-109X(19)30036-1. PMID 30879511
- [Derived] Kluyts HL, le Manach Y, Munlemvo DM, Madzimbamuto F, Basenero A, Coulibaly Y, Rakotoarison S, Gobin V, Samateh AL, Chaibou MS, Omigbodun AO, Amanor-Boadu SD, Tumukunde J, Madiba TE, Pearse RM, Biccard BM; African Surgical Outcomes Study (ASOS) investigators. The ASOS Surgical Risk Calculator: development and validation of a tool for identifying African surgical patients at risk of severe postoperative complications. Br J Anaesth. 2018 Dec;121(6):1357-1363. doi: 10.1016/j.bja.2018.08.005. Epub 2018 Sep 17. PMID 30442264
- [Derived] Biccard BM, Madiba TE, Kluyts HL, Munlemvo DM, Madzimbamuto FD, Basenero A, Gordon CS, Youssouf C, Rakotoarison SR, Gobin V, Samateh AL, Sani CM, Omigbodun AO, Amanor-Boadu SD, Tumukunde JT, Esterhuizen TM, Manach YL, Forget P, Elkhogia AM, Mehyaoui RM, Zoumeno E, Ndayisaba G, Ndasi H, Ndonga AKN, Ngumi ZWW, Patel UP, Ashebir DZ, Antwi-Kusi AAK, Mbwele B, Sama HD, Elfiky M, Fawzy MA, Pearse RM; African Surgical Outcomes Study (ASOS) investigators. Perioperative patient outcomes in the African Surgical Outcomes Study: a 7-day prospective observational cohort study. Lancet. 2018 Apr 21;391(10130):1589-1598. doi: 10.1016/S0140-6736(18)30001-1. Epub 2018 Jan 3. PMID 29306587
- See also: ASOS website — http://www.asos.org.za/
- Available data/document: Study Protocol — http://www.asos.org.za/ — ASOS Protocol version 1.0